CLINICAL TRIAL: NCT03321305
Title: Freshman Health Study
Brief Title: Eating Frequency and Visceral Adipose Tissue, Body Fat, and Obesity Risk in Hispanic College Freshmen
Acronym: FHS
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-11-0017
Record Dates: First submitted 2017-10-16; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Metabolic Disease; Eating Behavior; Adiposity; Sleep; Physical Activity
MeSH Terms: conditions — Obesity; Metabolic Diseases; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fasting Blood Draw: A fasting blood sample of four tablespoons will be obtained using a certified phlebotomist.
  Stool Sample: Participants will be instructed to collect the fecal sample wipe, which will then be stored in a labeled biosafety bag.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the increased focus on education and changing lifestyle, college students are particularly susceptible to poor overall health and wellness due to inadequate sleep and poor dietary choices. This is particularly important because the behavioral choices college students make may affect their risk of chronic disease. This study will research these topics via an online survey, in person visit and stool sample.

DETAILED DESCRIPTION:
It is important for college students to establish healthy habits during college because they are likely to stay with them throughout their lives. The transition to college has been identified as a critical period contributing to the rise in obesity rates. Several studies have shown that the initial transition to college is associated with rapid weight gain and the average weight gain in the first year of college ranges from 3.5 to 8.8 pounds. While decreased dietary fiber, fruits and vegetables and junk food consumption are among the dietary factors that have been linked to increased obesity rates in college students, little is known about the effect of eating patterns on health in this population. Furthermore, lack of sleep, smoking, binge drinking, and infrequent eating are all associated with negative health outcomes. Previous work with college age youth has found that several behaviors cluster together. The goal of the Online Survey portion is to expand on current findings, as well as examine the interrelationships of alcohol use, sleep, smoking, and eating patterns with adiposity and metabolic disease risk in a population of freshmen college students.

Eating frequency research has consistently found a negative association between the number of eating occasions (EOs) per day and adiposity, as well as metabolic disease risk in both youth and adult populations. Our group has shown that infrequent eating is linked to increased obesity measures, blunted insulin action, and deleterious lipid parameters in multiple populations of overweight Hispanic youth (8-18y). However, to date, no group has looked at the effect of eating frequency on adiposity and metabolic disease risk in a sample of overweight Hispanic college freshmen. In 2012, for the first time in history Hispanic high school graduates (69%) were more likely to be enrolled in college than Non-Hispanic Whites (NHW; 67%) and Blacks (63%) and last year Hispanic students represented 24% of freshman enrollment at the University of Texas at Austin (UT), Hispanics also showed the largest increase among all minority groups. Thus, the goal of the In-Person Visit is to examine the relationship between eating frequency and adiposity/metabolic disease risk in this extremely high-risk population of Hispanic freshmen and potentially identify interventions that may reduce this risk within such a crucial period of life.

The human body contains 100 trillion microbes, and microbial genes outnumber human genes 100:110. Over the past decade, interest in the complex ecosystem of gut microbiota has increased immensely and research has uncovered a relationship between gut microbiota, metabolic disease, and obesity. Both diet and obesity have been shown to alter the gut microbiota12,13. However, few studies have investigated how individual dietary components can affect the gut microbiota in humans. The Stool Sample portion of the study is an exploratory investigation of the relationship between dietary components and gut microbiota composition in college-aged Hispanic freshmen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Ages 18-24 years;
* Self-reported Hispanics (all four grandparents must be Hispanic)
* 50% of the sample will be self reported infrequent eaters (those who eat less than 2 eating occasions per day), as measured by 24-hr recalls
* 50% of the sample will be self-reported frequent eaters (those who report 3 or more eating occasions per day)
* A natural selection of normal, overweight and obese subjects will be recruited.

Exclusion Criteria:

* Subjects with serious medical disease as identified from a health history form;
* Pregnant;
* Taking any medications known to influence body composition or glucose/insulin action or psychoactive medications;
* Are diagnosed with diseases that may influence glucose/insulin indices or body composition;
* Have participated in a weight loss, dietary, or physical activity intervention in the past 6 months;
* Have a learning impairment that would complicate survey administration;
* Have braces, a pacemaker, or any other contraindications to MRI scanning, as visceral adipose tissue is a primary outcome

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For the survey portion of this study will be general in that participants must be currently enrolled freshmen students at UT Austin. Students can be male or female and of any ethnicity. Participants must be 18 years of age or older.
  The In-Person Visit inclusion/exclusion criteria will be more extensive and include the following:
  Ethnicity: This portion of the study will be limited to self-reported Hispanics because of their high risk of visceral adiposity and metabolic disorders.
  Eating Frequency We will enroll half Infrequent Eaters (≤2 EOs per day) and half Normal Eaters (≥3 EOs per day). Eating frequency groups will be identified via the previous survey data and verified with 24-hour diet recalls.
  BMI Status: We will include a natural selection of normal, overweight and obese students based on the Centers for Disease Control growth charts.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
College Students Habits and Obesity Risk | 2013-2017
  Examine the interrelationships of alcohol use, sleep, smoking, eating patterns, and physical activity with obesity (i.e., BMI parameters as measured by height in meters and weight in kilograms) in a population of freshmen college students
College student habits and type 2 diabetes risk factors | 2013-2017
  Examine the interrelationships of alcohol use, sleep, smoking, eating patterns, and physical activity with type 2 diabetes risk factors (i.e., glucose, insulin, insulin resistance as measured by fasting blood glucose) in a population of freshmen college students
College student habits and adiposity | 2013-2017
  Examine the interrelationship of alcohol use, sleep, smoking,eating patterns, and physical activity on adiposity (i.e., total body fat as measured by BodPod and visceral fat and liver fat as measured by MRI).

SECONDARY OUTCOMES:
Stool Samples and Gut Microbiome | 2013-2017
  Exploratory investigation of the relationship between dietary components and gut microbiota composition (specifically microbial diversity) in college-aged Hispanic freshmen
College Habits and Circulating lipids | 2013-2017
  Examine the interrelationship of alcohol use, sleep, smoking, eating patterns and physical activity levels on lipids (i.e., total cholesterol, triglycerides, and very low-density lipoprotein as measured by fasting blood draw).

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie N Davis, PhD,RD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared. Only aggregate data.